CLINICAL TRIAL: NCT00256256
Title: The Effect of GLP-1 on Glucose Uptake in the CNS and Heart in Healthy Subjects During Normoglycaemia Assessed by Positron Emission Tomografi
Brief Title: The Effect of GLP-1 on Glucose Uptake in the Brain and Heart in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2005-0079
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-10

CONDITIONS: Type 2 Diabetes; Stroke; Myocardial Infarction
Keywords: type 2 diabetes; GLP-1; PET; brain; heart
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Stroke; Myocardial Infarction | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: glucagon-like-peptide-1 — Dose: 1.2pmol/kg/min for 6 hours

SUMMARY:
Type 2 diabetes mellitus, T2D is a disease characterized by an immense growing prevalence world wide with an increased risk of myocardial infarction and stroke. GLP-1 has convincing effects on the high glucose levels in type 2 diabetic patients and is well tolerated. New animal studies indicate a protective effect of GLP-1 in the brain and the heart. The mechanism behind this is yet not known.

The study hypothesis is that GLP-1 will stimulate glucose-uptake in the brain and heart independent of insulin and thereby exert its protective effects.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus, T2D is a disease characterized by an immense growing prevalence world wide. T2D is associated with a three-fold increase in cardiovascular complications (myocardial infarction and stroke) leading to significantly higher morbidity and mortality in this group of patients. The prospective British Diabetes Study (UKPDS) showed that neither diet alone nor the pharmaceutical treatment utilized (Sulphonylurea, Metformin, Insulin) were able to reduce these macrovascular complications. GLP-1 (glucagon-like-peptide-1)is an incretin with convincing effects on glycaemia in type 2 diabetic patients with little or no risk of hypoglycaemia. New research in animal models has shown a potential protective effect in the brain and heart in association with ischaemic damage. The mechanism behind this protective effect is not known.

The effect of native GLP-1 on glucose uptake in the brain and heart will by visualized by fluoro-deoxy-glucose FDG-PET-scan during normoglycaemia in healthy young men. At the same time a pancreatic/pituitary clamp will be performed. The hypothesis is that GLP-1 directly will stimulate glucose uptake independent of the pancreatic hormones and through this mechanism exert its neuro- and cardioprotective actions.

Comparisons: FDG-uptake in the brain and heart with GLP-1 infusion compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Age 20-50 years
* Caucasian
* BMI 20-30 kg/m2

Exclusion Criteria:

* Diabetes in subject and 1.degree relatives
* Any disease of clinical relevance

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-11; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
FDG-uptake in the brain and heart visualized by Positron emission tomography with and without GLP-1 | After 4 hours of GLP-infusion

SECONDARY OUTCOMES:
Laboratory values (insulin secretion and counter-regulatory hormones) | During 7 hours of clamp and GLP-1/placebo infusion

CONTACTS AND LOCATIONS:
Overall Officials: Ole Schmitz, MD,professor, Principal Investigator — Department of pharmacology, Aarhus university
Locations (1):
- Department of pharmacology, Aarhus university, Aarhus, Denmark

REFERENCES:
- [Background] During MJ, Cao L, Zuzga DS, Francis JS, Fitzsimons HL, Jiao X, Bland RJ, Klugmann M, Banks WA, Drucker DJ, Haile CN. Glucagon-like peptide-1 receptor is involved in learning and neuroprotection. Nat Med. 2003 Sep;9(9):1173-9. doi: 10.1038/nm919. Epub 2003 Aug 17. PMID 12925848
- [Background] Nikolaidis LA, Mankad S, Sokos GG, Miske G, Shah A, Elahi D, Shannon RP. Effects of glucagon-like peptide-1 in patients with acute myocardial infarction and left ventricular dysfunction after successful reperfusion. Circulation. 2004 Mar 2;109(8):962-5. doi: 10.1161/01.CIR.0000120505.91348.58. Epub 2004 Feb 23. PMID 14981009
- [Background] Holst JJ. On the physiology of GIP and GLP-1. Horm Metab Res. 2004 Nov-Dec;36(11-12):747-54. doi: 10.1055/s-2004-826158. PMID 15655703
- [Background] Perry T, Haughey NJ, Mattson MP, Egan JM, Greig NH. Protection and reversal of excitotoxic neuronal damage by glucagon-like peptide-1 and exendin-4. J Pharmacol Exp Ther. 2002 Sep;302(3):881-8. doi: 10.1124/jpet.102.037481. PMID 12183643
- [Background] Bose AK, Mocanu MM, Carr RD, Yellon DM. Glucagon like peptide-1 is protective against myocardial ischemia/reperfusion injury when given either as a preconditioning mimetic or at reperfusion in an isolated rat heart model. Cardiovasc Drugs Ther. 2005 Jan;19(1):9-11. doi: 10.1007/s10557-005-6892-4. No abstract available. PMID 15883751
- [Derived] Gejl M, Lerche S, Mengel A, Moller N, Bibby BM, Smidt K, Brock B, Sondergaard H, Botker HE, Gjedde A, Holst JJ, Hansen SB, Rungby J. Influence of GLP-1 on myocardial glucose metabolism in healthy men during normo- or hypoglycemia. PLoS One. 2014 Jan 6;9(1):e83758. doi: 10.1371/journal.pone.0083758. eCollection 2014. PMID 24400077